CLINICAL TRIAL: NCT06281964
Title: Randomized, Controlled, Open Label, Multicenter Phase III Study to Evaluate the Efficacy and Safety of PLB1004 Versus Platinum-based Chemotherapy With or Without Sintilimab of Advanced NSCLC With EGFR Exon 20 Ins Mutations
Brief Title: Efficacy and Safety Evaluation of PLB1004 in Patients With Non-squamous NSCLC Harboring EGFR Exon 20 Insertion.
Acronym: KANNON-2
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Avistone Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PLB1004-III-01
Record Dates: First submitted 2024-01-31; First posted 2024-02-28 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Non-Small-Cell Lung Cancer
Keywords: Non-Small-Cell Lung Cancer; EGFR; NSCLC; Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PLB1004 (Experimental): PLB1004 given alone as monotherapy
  Interventions: Drug: PLB1004
- platinum-based chemotherapy with or without Sintilimab (Active Comparator): platinum-based chemotherapy with or without Sintilimab
  Interventions: Drug: Pemetrexed+（carboplatin or Cisplatin）with or without Sintilimab

INTERVENTIONS:
Drug: PLB1004 — Participants received oral PLB1004 240mg on Day 1 every 3 weeks (q3w), IV infusion of 500 milligrams per meter square (mg/m^2) pemetrexed on Day 1 q3w, and as per investigator's choice either IV infusion of carboplatin on Day 1 q3w with a dose calculated using 'Calvert formula' to obtain area under concentration versus time (AUC) = 5 milligrams per milliliter per minute (mg/mL/min) or IV infusion of 75 mg/m^2 cisplatin q3w on Day 1 q3w, during induction dosing period of 4 or 6 cycles (Cycle length=21 days). Participants who experienced clinical benefit during the induction phase began maintenance therapy. Participants will receive oral PLB1004 240mg and 500 mg/m^2 of pemetrexed on Day 1 q3w until disease progression in the maintenance period.
  Arms: PLB1004
Drug: Pemetrexed+（carboplatin or Cisplatin）with or without Sintilimab — Participants received IV infusion of 500 milligrams per meter square (mg/m^2) pemetrexed on Day 1 q3w, and as per investigator's choice either IV infusion of carboplatin on Day 1 q3w with a dose calculated using 'Calvert formula' to obtain area under concentration versus time (AUC) = 5 milligrams per milliliter per minute (mg/mL/min) or IV infusion of 75 mg/m^2 cisplatin q3w on Day 1 q3w, during induction dosing period of 4 or 6 cycles (Cycle length=21 days). Sintilimab 200mg intravenously administered on day 1 q3w per investigator's decision. Participants who experienced clinical benefit during the induction phase began maintenance therapy. Participants will receive oral PLB1004 and 500 mg/m^2 of pemetrexed on Day 1 q3w and Sintilimab 200mg intravenously administered on day 1 q3w per investigator's decision. until disease progression in the maintenance period.
  Arms: platinum-based chemotherapy with or without Sintilimab

SUMMARY:
Efficacy and safety evaluation of PLB1004 in patients with locally advanced/metastatic non-squamous NSCLCharboring EGFR exon 20 insertion.

DETAILED DESCRIPTION:
Randomized, controlled, open label, multicenter phase III study to evaluate the efficacy and safety of PLB1004 Versus platinum-based chemotherapy with or without Sintilimab in the first-line treatment of locally advanced or metastatic non-squamous non-small cell lung cancer with Epidermal Growth Factor Receptor (EGFR) Exon 20 insertion(ex 20) mutations.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and willingness to sign a written informed consent document.
2. Aged at least 18 years old.
3. Histologically or cytologically confirmed locally advanced or metastatic NSCLC (stage IIIB~IV).
4. Tumor tissue is positive for EGFR Ex20ins as documentally confirmed by next-generation sequencing (NGS) testing or written confirmation of PCR testing by a local laboratory accredited by the Clinical Laboratory Improvement Act Amendments (CLIA), International Organization for Standardization/Independent Ethics Committee (ISO/IEC), American College of Pathologists (CAP), or a central laboratory designated by the sponsor by a tertiary A hospital or with Clinical Laboratory Improvement Act Amendments (CLIA), International Organization for Standardization/Independent Ethics Committee (ISO/IEC), American College of Pathologists (CAP) accreditation (or other equivalent accreditation).
5. At least one measurable lesion as defined by RECISTV1.1（Brain lesions were not included in measurable target lesions）
6. ECOG performance status 0 to 1.
7. Life expectancy is not less than 12 weeks.
8. No previous systemic treatment for locally advanced or metastatic non-squamous cell cancer NSCLC. Note: Subjects are allowed to receive neoadjuvant/adjuvant therapy as long as the relevant therapy has ended at least 6 months before the disease is diagnosed as locally progressive or metastatic tumors

   -

Exclusion Criteria:

1. Have one of the following previous anti-tumor treatments: prior to the first dose of PLB1004

   a) Any anti-EGFR TKI for the EGFR ex20ins mutation.. b) Received Chinese patent drugs with anti-tumor indications within 1 week before administration of the first study drugReceived Chinese patent drugs with anti-tumor indications within 1 week before administration of the first study drug c) required administration of the multidrug and toxin efflux protein (MATE) transporter substrate metformin within 1 week before and during the first study drug administration d）Strong inhibitors or strong inducers of the cytochrome P450 3A4 enzyme (CYP3A4) were required within 1 week before and during the study e) required immunosuppressive medication within 2 weeks before or during the first dose of study drug f) Major surgery within 4 weeks prior to starting PLB1004 or who have not recovered from side effects of such procedure except for the biopsy of Thoracoscopy and the clinical test of Mediastinoscopy could ≤ 7 days prior to starting PLB1004 g) Radiotherapy to lung fields and whole-brain fields ≤4 weeks prior to starting PLB1004. For all other anatomic sites, radiotherapy ≤2 weeks prior to starting PLB1004 or patients who have not recovered from radiotherapy-related toxicities. Palliative radiotherapy for bone lesions is not included.
2. Patients with spinal cord compression ,brain membrane metastasis and symptomatic central nervous system (CNS), who are neurologically unstable or have required increasing doses of steroids within the 2 weeks prior to study manage CNS symptoms.
3. Before randomization, patients did not recover from any toxicity and/or complications of previous chemotherapy, surgery, radiotherapy and other anti-cancer treatments, that is, did not fall to grade 1 or lower (National Cancer Research Common Toxicity Criteria for Adverse Events [NCI-CTCAE] v5.0), except for hair loss and irrecoverable permanent radiation damage
4. Did not recover from any toxicity and/or complications of previous anti-cancer treatments such as chemotherapy, surgery, and radiotherapy, that is, did not fall to grade 1 or lower (National Cancer Research Common Toxicity Criteria for Adverse Events [NCI-CTCAE] v5.0), except for alopecia and irrecoverable permanent radiation damage
5. A tendency to coagulopathy or bleeding, including an arterial or venous thromboembolic event (including a history of myocardial infarction, unstable angina, cerebrovascular accident or transient ischemic attack, pulmonary embolism, deep vein thrombosis, or any other major thromboembolism) within 6 months before randomization; Any life-threatening bleeding event (including the need for blood transfusion, surgical or local treatment, or continued medical therapy) or major vascular invasion was considered by the investigator to be bleeding prone
6. Severe cardiac disease, such as any serious arrhythmia (including ventricular arrhythmia, drug-refractory supraventricular and other arrhythmias), grade III or higher cardiac dysfunction (New York Heart Association [NYHA], see Appendix 4 for details), and left ventricular ejection fraction (LVEF) <50% on echocardiography;
7. Mean corrected QT intervals (QTcF) of three electrocardiograms during screening, calculated according to Fridericia's formula at rest, were >470 ms;
8. Presence of uncontrolled hypertension (treated systolic blood pressure >160 mmHg and/or diastolic blood pressure >100 mmHg)
9. Dysphagia, or active digestive disease or major gastrointestinal surgery that may affect the administration or absorption of the study drug (e.g., ulcerative lesions, uncontrolled nausea, vomiting, diarrhea, and malabsorption syndromes);
10. Allergy or intolerance to the drug class and excipient components of the study drug
11. pregnant or nursing women.
12. Received live vaccine within 4 weeks before randomization;

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) by BICR | 3 years
  Progression-free survival (PFS) as assessed by a Blind Independent Center Review Committee (BICR) with reference to RECIST v1.1 for Solid tumors

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) by the investigator | 2 years
  Refer to RECIST v1.1, PFS assessed by the investigator
Intracranial Overall Response Rate（ORR） | 3 years
  To evaluate the intracranial Overall Response Rate（ORR）which is defined by investigator as the proportion of subjects with Intracranial disease confirmed best overall response of complete response or partial response per RECIST v 1.1.
Duration of Response (DOR) | 3 years
  DOR is defined as the time from the date of first documented response (CR or PR) until the date of documented progression or death, whichever comes first.
Disease Control Rate (DCR) | 3 years
  DCR is defined as the percentage of participants achieving complete or partial response or stable disease as defined per RECIST v 1.1
Overall Survival (OS) | 3 years
  OS is defined as the time from the date of the first dose until the date of death due to any cause.
Incidence of Treatment-Emergent Adverse Events (TEAEs) | 3 years
  A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug assessed by CTCAE v5.0
Plasma concentrations of PLB1004 and metabolites may be combined with data from other clinical studies | 3 years
  Plasma concentrations of PLB1004 and metabolites may be combined with data from other clinical studies

OTHER OUTCOMES:
intracranial Progression-Free Survival（PFS） | 3 years
  Reference RECIST v1.1, intracranial PFS assessed by BICR and investigator
Time to second progression-free survival(PFS2) | 3 years
  Time to second progression-free survival (PFS2) as assessed by the investigator
Assess the Quality of Healthy Living About Patients | 3 years
  Use the EQ-5D-5L scale to measure patients' quality of healthy living. It has 5 items (Mobility, Self-care, Usual activities, Pain/discomfort, Depression/anxiety). Each item contains 5 levels: 1= no difficulty, 2= slight difficulty, 3= moderate difficulty, 4= serious difficulty, 5= extremely serious difficulty. The higher the score has the worse the health. Then, the score calculation of the European Five-Dimensional Health Scale is based on the calculation formula published by the EuroQol Group. Based on 5 combinations of different severity levels, a score of 0 to 1 is obtained. 0 is the least healthy and 1 is the most healthy.
EGFR Ex20ins status in tumor tissues and its relevance to the clinical efficacy of drugs | 3 years
  EGFR Ex20ins status in tumor tissues and its relevance to the clinical efficacy of drugs
Gene mutation status in plasma ctDNA before and after medication, and its correlation with clinical efficacy | 3 years
  To assess the expression of circulating tumor DNA in ascites and blood, ctDNA was mesured at screen, cycle 3 and end of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No